CLINICAL TRIAL: NCT03194230
Title: Interest of Cervical Dilators in the Induction of Labor in Second Trimester Medical Termination of Pregnancy.
Brief Title: Interest of Cervical Dilators in Second Trimester Termination of Pregnancy
Acronym: DILATOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P160908
Record Dates: First submitted 2017-06-13; First posted 2017-06-21 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Termination of Pregnancy (TOP)
Keywords: Cervical dilators; induction of labor; cervical ripening; medical termination of pregnancy; second-trimester of pregnancy.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Without cervical dilator (No Intervention): Induction of labour by oral of 400µg of misoprostol each 3 hours.
- With cervical dilator (Experimental): Induction of labour by cervical placement of hygroscopic dilators for 3 hours and oral of 400µg tablets of misoprostol each 3 hours.
  Interventions: Other: With cervical dilatator

INTERVENTIONS:
Other: With cervical dilatator — Induction of labour by cervical placement of hygroscopic dilators (Dilapan-S Hygroscopic cervical dilator )
  Arms: With cervical dilator

SUMMARY:
The purpose of this study is to evaluate whether the use of cervical dilators for cervical ripening in case of second trimester medical termination of pregnancy (TOP) is effective to reduce duration of labor.

DETAILED DESCRIPTION:
Termination of pregnancy is a distressing and painful procedure for women. The use of cervical dilators could shorten the duration of labor but can generate more pain. The investigators will compare two procedures of induction of labor for second trimester termination of pregnancy: one with the use of oral prostaglandins (misoprostol) only and one with the exact same procedure preceded by cervical ripening with hygroscopic cervical dilators. Epidural analgesia will be effective previously to the placement of cervical dilators and the first tablet of misoprostol. Efficacy will be determined based on the proportion of women achieving vaginal delivery within 12 hours. The beginning of labor will be defined as the first administration of misoprostol tablets in both groups.

The investigators will also evaluate safety by collecting hemorrhage endometritis, cervical tear. The investigators will compare psychological impact of these procedures, measured by the impact of event scale and acceptability 1 to 4 months later.

ELIGIBILITY:
Inclusion Criteria:

* Termination of pregnancy requested by the patient and accepted by the weekly multidisciplinary counselling of fetal medicine
* gestational age between 15 and 27 weeks and 6 days,
* single pregnancy,
* major patient,
* French-speaking woman,
* Patient with health insurance.

Exclusion Criteria:

* Termination of pregnancy by surgical technique
* cicatricial uterus
* premature rupture of membranes
* chorioamnionitis
* multiple pregnancy
* placenta praevia
* myoma praevia
* uterine malformation
* unstable maternal pathology
* psychiatric pathology
* contraindication to mifepristone: severe asthma, adrenal insufficiency, porphyria, corticotherapy.
* contraindication to misoprostol: hypersensitivity to prostaglandins.
* contraindication to epidural analgesia: hemostasis disorder, spinal or medullary anomaly.
* Bishop score > or = to 7 at arrival in birth room

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Proportion of women achieving vaginal delivery within 12 hours | 12 hours
  The beginning of labor will be defined as the placement of the first tablets of misoprostol in both groups.

SECONDARY OUTCOMES:
Induction-to-amniotomy interval | 12 hours
  Time between the first placement of misoprostol tablets and artificial amniotomy.
Induction-to-delivery interval | 24 hours
  Time between the first placement of misoprostol tablets and delivery.
Failure in induction of labor | 24 hours
  Proportion of women not achieving vaginal delivery within 24 hours
Pain assessment at the beginning of the procedure | Hour 0
  Pain assessment with numerical scale at the placement of dilators and the first misoprostol tablets
Pain assessment of the whole procedure of TOP | 48 hours
  Pain assessment of the whole procedure by numerical scale at discharge of the hospital
Distress assessment at discharge after TOP | 4 months
  Distress assessment at discharge after TOP measured by impact of event scale revised(IES-R)
Assessment of acceptability of the whole procedure of TOP | 4 months
  Acceptability measured by the proportion of women who would opt for the same procedure after TOP
number of complications. | 4 months
  Hyperthermia> 40 ° C, septicemia, endometritis defined by a fever associated with pelvic pain, positive bacteriological vaginal specimen and a biological infectious syndrome (leukocytosis greater than 15 000 / mm3 and C-Reactive Protein > 10 IU / mL).
  * Cervical injury.
  * Complications of prolonged decubitus: bedsores, thrombo-embolic complications.
  * Uterine rupture.
  * Post-partum hemorrhage defined by estimated blood losses greater than 500 mL.
Duration of hospitalization. | 48 hours
  Duration of hospitalization between admission and discharge and in delivery room.
Cost of the procedure | 4 months
  Assessment of the whole procedure costs of TOP, including potential complications.
Among nullipara, proportion of women achieving vaginal delivery within 12 hours | 12 hours
  The beginning of labor will be defined as the placement of the first tablets of misoprostol in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Tsatsaris, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Maternité Port Royal, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anselem O, Jouannic JM, Winer N, Bouchghoul H, Vivanti AJ, Quibel T, Massardier J, Rousseau J, Ancel PY, Goffinet F, Tsatsaris V. Cervical Dilators Used Concurrently With Misoprostol to Shorten Labor in Second-Trimester Termination of Pregnancy: A Randomized Controlled Trial. Obstet Gynecol. 2022 Sep 1;140(3):453-460. doi: 10.1097/AOG.0000000000004887. Epub 2022 Aug 3. PMID 35926202
- [Background] Vincienne M, Anselem O, Cordier AG, Le Ray C, Tsatsaris V, Benachi A, Goffinet F. Comparison of the Induction-to-Delivery Interval in Terminations of Pregnancy with or without Dilapan-S(R). Fetal Diagn Ther. 2018;43(1):61-67. doi: 10.1159/000458410. Epub 2017 Mar 29. PMID 28351055
- [Background] Jain JK, Mishell DR Jr. A comparison of misoprostol with and without laminaria tents for induction of second-trimester abortion. Am J Obstet Gynecol. 1996 Jul;175(1):173-7. doi: 10.1016/s0002-9378(96)70270-3. PMID 8694046
- [Background] Mazouni C, Vejux N, Menard JP, Bruno A, Boubli L, d'Ercole C, Bretelle F. Cervical preparation with laminaria tents improves induction-to-delivery interval in second- and third-trimester medical termination of pregnancy. Contraception. 2009 Jul;80(1):101-4. doi: 10.1016/j.contraception.2009.01.013. Epub 2009 Mar 4. PMID 19501224
- [Background] Pluchon M, Winer N. [Misoprostol in case of termination of pregnancy in the second and third trimesters. Trials]. J Gynecol Obstet Biol Reprod (Paris). 2014 Feb;43(2):162-8. doi: 10.1016/j.jgyn.2013.11.009. Epub 2014 Jan 16. French. PMID 24440001
- [Background] Gitz L, Morel O, Thiebaugeorges O, Sibiude J, Desfeux P, Barranger E. [Termination of pregnancy and intra-uterine fetal death after 14 weeks of pregnancy: Which protocol for induction of labour in 2010?]. J Gynecol Obstet Biol Reprod (Paris). 2011 Feb;40(1):1-9. doi: 10.1016/j.jgyn.2010.11.007. Epub 2010 Dec 23. French. PMID 21185133
- [Background] Thong KJ, Baird DT. A study of gemeprost alone, dilapan or mifepristone in combination with gemeprost for the termination of second trimester pregnancy. Contraception. 1992 Jul;46(1):11-7. doi: 10.1016/0010-7824(92)90127-f. PMID 1424619